CLINICAL TRIAL: NCT03041194
Title: Title A Pilot Study to Evaluate the Dietary Impact on Urinary pH in Interstitial Cystitis Pilot Study to Evaluate the Dietary Impact on Urinary pH in Interstitial Cystitis
Brief Title: Dietary Impact on Urinary pH in Women With Interstitial Cystitis
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Rosemary Catanzaro, RD, Principal Investigator, St. Louis University
Other Study IDs: 25300
Record Dates: First submitted 2017-01-19; First posted 2017-02-02 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: dietary affects — Dietary affects on urine pH in relation to Interstitial cystitis symptoms

SUMMARY:
This is a pilot study on subjects who suffer from Interstitial Cystitis (IC) to assess the dietary affects on urine pH in relation to their symptoms. The goal of this pilot study is to determine which foods/beverages affect urinary pH and exacerbate patient's symptoms.

DETAILED DESCRIPTION:
Interstitial cystitis or painful bladder syndrome is a condition that is chronic and often debilitating in nature. Interstitial cystitis is commonly defined by symptoms of urinary urgency and frequency associated with pelvic pain. Around one million men and women in the United States and Europe suffer from this condition. The diagnosis of Interstitial Cystitis is one of exclusion based on cystoscopy findings and clinical symptoms. Common symptoms of Interstitial Cystitis include urinary frequency, urinary urgency, dysuria, and pain in the lower abdominal region, bladder, vagina, urethra, or in the perinea . Women between ages 40 and 60 are the most commonly affect by Interstitial Cystitis. In the Nurses' Healthy Study I and II the prevalence of Interstitial Cystitis was 52-67 individuals out of 100,000. There is no single cause of Interstitial Cystitis however, there are several known theories to the cause of Interstitial Cystitis. A popular hypothesis is that a defect in the glycosaminoglycan layer of the bladder epithelium allows leakage and absorption of urinary solutes. The major solute that is responsible for causing bladder symptoms when the epithelium is injured is potassium. The long held notion is that patients with Interstitial Cystitis should avoid acidic foods. This logic is largely based on anecdotal data and questionnaires of foods, beverages and supplements that increase symptoms. Controversy exists that Interstitial Cystitis diet restricts many more foods than necessary in an attempt to decrease Interstitial Cystitis symptoms. Current questionnaires-based data suggest eliminating tomatoes, citrus fruits, vitamin C, artificial sweeteners, carbonated and alcoholic beverages, and spicy foods which are thought to exacerbate symptoms, while calcium glycerophosphate and sodium bicarbonate may improve symptoms. Though the literature review, the investigators did not find any analytical studies that correlated diet with Interstitial Cystitis symptoms or that the ingestion of acidic foods exacerbate Interstitial Cystitis symptoms. Based on the lack of analytical data and the impact of acidic food on IC symptoms this study is going to evaluate the potential renal acid load and net acid excretion of foods to determine which foods change urinary pH.

ELIGIBILITY:
Inclusion Criteria:

* Women, diagnosed with Interstitial Cystitis or with a presumptive clinical diagnosis of IC
* New IC patients who agree to hydrodistention and cystoscopy, the standard of care for diagnosis of IC

Exclusion Criteria:

* Subjects who are diagnosed with Fibromyalgia Syndrome and subjects that are pregnant.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female, all backgrounds and races
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The impact of urinary pH | 1 year
  urinary pH.

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Catanzaro, MS RD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No